CLINICAL TRIAL: NCT06257784
Title: Single Breath Counting Test for Acute Respiratory Failure in Emergency Department: Multicenter Observational Prospective Trial (STARED-TRIAL)
Brief Title: Single Breath Counting Test for Acute Respiratory Failure in Emergency Department
Acronym: STARED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.RianGen.22.01
Record Dates: First submitted 2023-05-11; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Failure
Keywords: Single breath counting test; Acute Respiratory Failure
MeSH Terms: interventions — Oxygen; Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Respiratory Failure: Every patient admitted in Emergency department with any acute respiratory failure will be screened according to inclusion and exclusion criteria to being recruited in the study
  Interventions: Procedure: Oxygen Therapy; Procedure: Non-Invasive Ventilation (NIV); Procedure: Invasive Ventilation

INTERVENTIONS:
Procedure: Oxygen Therapy — Patients who have SpO2 < 92% on room air will undergo oxygen therapy (nasal cannula or Venturi-mask).
Procedure: Non-Invasive Ventilation (NIV) — Patients with P/F < 250 or Ph < 7,35 with PCO2 > 50 mmHg will undergo Non-Invasive Ventilation (NIV) (high flow nasal cannula or CPAP).
Procedure: Invasive Ventilation — Patients with P/F < 150 associated to dyspnea at rest (moderate to severe, shortness of breath and/ or tachypnea (>24 breaths/min) despite NIV for at least 2 hours or patients with Ph < 7,2 with PCO2 > 60 mmHg despite NIV for at least 2 hours will undergo invasive ventilation (intubation).

SUMMARY:
The purpose of the study is to determine whether SBCT is a useful tool for diagnosing the main form of failure respiratory acute and to define the SBCT limit associated with insufficiency respiratory in this population, the requirement for NIV or invasive ventilation.

Furthermore, the correlation with the most common scores and indices used in the emergency room will be studied, such as: HACOR, MEW, REMS SCORE, ROS, CURB-65, qSOFA, SEVERITY INDEX OF PNEUMONIA, GWTG HF, LUNG ULTRASOUND SCORE, SINGLE BREATH COUNT

DETAILED DESCRIPTION:
Single breath counting test (SBCT) is the measurement of how far an individual can count in a normal speaking voice after a maximal effort inspiration. Previous work has demonstrated that SBCT has good correlation with the gold standard measures of pulmonary function test, peak expiratory flow rate and forced expiratory volume in the first second.

The easy of the SBCT makes this test appealing for rapid assessment of respiratory status overall in patients admitted for acute respiratory failure and we hypothesized that it will be valuable, replicable and fast tools for bedside assessment of respiratory function in Emergency Department.

The purpose of the study is to determine whether SBCT is a useful tool for diagnosis of the major form of acute respiratory failure and to define the cut-off limit of SBCT associated to respiratory failure in this population, requirement of NIV or invasive ventilation. Moreover, it will be studied the correlation with the most common scores and indexes used in emergency department like: HACOR, MEW, REMS SCORE, ROS, CURB-65, qSOFA, PNEUMONIA SEVERITY INDEX, GWTG-HF, LUNG ULTRASOUND SCORE, SINGLE BREATH COUNTING TEST

ELIGIBILITY:
Inclusion Criteria:

* Any Acute Respiratory Failure
* SaO2 <92% on air room at ED admission

Exclusion Criteria:

* Age < 18 yo
* Patients already in NIV AND HCFN in ED
* Home-oxygen or Home-NIV therapy
* SpO2 < 80%
* Severe dyspnea
* unable to speak complete sentences
* Uncooperative patients
* Hemodynamic Instability < 90 mmHg or vasopressor requirement at admission
* ST Elevation-Miocardial Infarction
* Tracheo -stomized or -tomized patients
* End of life

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with any Acute Respiratory Failure admitted in Emergency department
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Single Breath Counting Test (SBCT) | Change from Baseline at 3 hours
  Determine if SBCT is a useful, fast and reproducible tool for assessing respiratory failure and its severity in the Emergency Department.

SECONDARY OUTCOMES:
SBCT as predictor NIRS | Change from Baseline at 3 hours
  Define if Single Breath Counting Test (SBCT) could be a predictor of Non-Invasive Respiratory Strategies (NIRS)
Correlation with the main critical illness scores | Change from Baseline at 3 hours
  Define the correlation of SBCT with the main critical illness scores
Correlation with the main serum markers | Change from Baseline at 3 hours
  Define the correlation of SBCT with the main serum markers corresponding to the underlying respiratory failure disorder
Correlation with imaging | Change from Baseline at 3 hours
  Define the correlation of SBCT with radiographic (infiltrated) and ultrasound imaging
Cut-off limit of SBCT | Change from Baseline at 3 hours
  Define the cut-off limit, the sensitivity and the specificity of SBCT associated with respiratory failure
Cut-off limit to initiate appropriate respiratory support | Change from Baseline at 3 hours
  Define the cut-off limit to initiate appropriate respiratory support
Correlation with Emergency Room Mortality | Change from Baseline at 3 hours
  Define the correlation of SBCT with Emergency Room Mortality
Correlation between pulmonary and extrapulmonary causes | Change from Baseline at 3 hours
  Correlation between pulmonary and extrapulmonary causes

CONTACTS AND LOCATIONS:
Overall Officials: Yaroslava Longhitano, Physician, Principal Investigator — Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo
Locations (1):
- Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No